CLINICAL TRIAL: NCT01393977
Title: Efficacy Difference Between Rehabilitation Therapy and Umbilical Cord Derived Mesenchymal Stem Cells Transplantation in Patients With Acute or Chronic Spinal Cord Injury in China
Brief Title: Difference Between Rehabilitation Therapy and Stem Cells Transplantation in Patients With Spinal Cord Injury in China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2011-01-19SCI
Record Dates: First submitted 2011-07-06; First posted 2011-07-14 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Stem Cell Transplantation; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (No Intervention): Outpatient in hospital
- rehabilitation (Active Comparator): interventions: rehabilitation
  Interventions: Procedure: rehabilitation of limb function
- Stem Cell Transplantation (Experimental): interventions: stem cell transplantation
  Interventions: Procedure: Stem Cells Transplantation

INTERVENTIONS:
Procedure: rehabilitation of limb function — only receive rehabilitation of limb function
  Other Names: phsical exercise rehabilitation
  Arms: rehabilitation
Procedure: Stem Cells Transplantation — mesenchymal stem cells derived from umbilical cord are transplanted directly into subarachnoid by Lumbar puncture
  Arms: Stem Cell Transplantation

SUMMARY:
The morbidity of spinal cord injury (SCI) is increasing significantly in China. The methods to treat SCI patients in sequela stage update are poor. Though traditional rehabilitation therapy is the routine method to treat SCI in sequela stage, its effect to improve the neurological disorders of these patients, such as the dysfunction of sense, motor, autologous adjustment of blood pressure control of urination and defecation, perspiration , etc. is unsatisfying. Rehabilitation Therapy can prevent the process of muscle atrophy and joint stiffness. However, it can not repair the damaged nerve function. Studies show that mesenchymal stem cell transplantation can remarkably improve the neurological function of SCI in animals without any severe side effect.

In this study, the investigators use mesenchymal stem cells derived from umbilical cord to treat 40 SCI patients (20 cases in early stage and 20 cases in sequela stage). The investigators also follow-up ten patients who only receive rehabilitation and another ten outpatients who accept neither stem cell therapy nor rehabilitation. On this basis, the investigators can compare the efficacy of these two treatments.

DETAILED DESCRIPTION:
Patients enrolled in this study need to finish our whole follow-up survey, which is carried out by clinical doctors and epidemiologist.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their curator must be able to give voluntary consent.
2. Patients or their curator Must be able to understand the information of study and in which group they are.
3. 20 years - 50 years of age can be enrolled.
4. Both male and female can be enrolled.
5. Patients have clear history of traumatic injury, and the spinal cord injury are confirmed by all of the examinations including MRI, electromyogram and electrophysiology.

Exclusion Criteria:

1. Mental disorders
2. Myelitis
3. Women in pregnancy
4. Cancer

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Electromyogram and Electroneurophysiologic test | 3 monthes after enrollment or transplantation
  Brain stem auditory evoked potential (BAEP)and electromyography can display the nerve conduction velocity and the improvement of neurological function.

SECONDARY OUTCOMES:
Electromyogram and Electroneurophysiologic test | 6monthes after enrollment or transplantation
  Brain stem auditory evoked potential (BAEP)and electromyography can display the nerve conduction velocity and the improvement of neurological function.
Electromyogram and Electroneurophysiologic test | 12monthes after enrollment or transplantation
  Brain stem auditory evoked potential (BAEP)and electromyography can display the nerve conduction velocity and the improvement of neurological function.

CONTACTS AND LOCATIONS:
Overall Officials: An Yihua, doctor, Study Director — Chinese People's Armed Police Force
Locations (1):
- Yihua An, Beijing, China

REFERENCES:
- [Derived] Cheng H, Liu X, Hua R, Dai G, Wang X, Gao J, An Y. Clinical observation of umbilical cord mesenchymal stem cell transplantation in treatment for sequelae of thoracolumbar spinal cord injury. J Transl Med. 2014 Sep 12;12:253. doi: 10.1186/s12967-014-0253-7. PMID 25209445